CLINICAL TRIAL: NCT00715611
Title: Phase II Toxicity Study of Pleurectomy/Decortication, (Neo) Adjuvant Chemotherapy and Intensity Modulated Radiation Therapy to the Pleura in Patients With Locally Advanced Malignant Pleural Mesothelioma
Brief Title: Pleurectomy/Decortication (Neo) Adjuvant Chemotherapy and Intensity Modulated Radiation Therapy to the Pleura in Patients With Locally Advanced Malignant Pleural Mesothelioma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Princess Margaret Hospital, Canada (Other); Mayo Clinic (Other); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-053
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Mesothelioma
Keywords: pemetrexed; cisplatin; IMRT; PLEURA; Malignant; 08-053
MeSH Terms: conditions — Mesothelioma | interventions — Cerebral Decortication; Pemetrexed; Cisplatin; Carboplatin; Radiotherapy, Intensity-Modulated

ARMS (1):
- 1 (Experimental): This is a multicenter phase II toxicity study of pleurectomy/decortication (P/D) followed by adjuvant chemotherapy and Intensity Modulated Radiation Therapy (IMRT) to the pleura in patients with malignant pleural mesothelioma. Alternatively, chemotherapy may be administered in the neoadjuvant setting prior to P/D, followed by IMRT. Patients deemed resectable at the time of enrollment will undergo P/D with the goal of a macroscopic complete resection (MCR). Those with disease progression or severe toxicity will stop chemotherapy and undergo a PET scan.
  Interventions: Procedure: Pleurectomy/Decortication; Drug: pemetrexed and cisplatin or carboplatin; Radiation: Intensity Modulated Radiation Therapy

INTERVENTIONS:
Procedure: Pleurectomy/Decortication — Pleurectomy/decortication will be performed as per standard technique
  Other Names: (P/D)
Drug: pemetrexed and cisplatin or carboplatin — The combination of pemetrexed and cisplatin or carboplatin will be given every 3 weeks for up to 4 cycles. Pemetrexed will be administered at 500mg/m2 as a 10-minute infusion. Cisplatin will be administered at 75mg/m2 as a 60-minute infusion. Carboplatin will be administered at an AUC of 5 over 30 minutes. Chemotherapy may be administered in the neoadjuvant or adjuvant setting.
Radiation: Intensity Modulated Radiation Therapy — IMRT will be administered over approximately 6 weeks at 50.4 Gy in 28 fractions with an optional SIB to gross residual disease (pending meeting normal tissue constraints).
  Other Names: IMRT

SUMMARY:
For patients with this type of cancer, the standard of care is treatment with chemotherapy. Radiation therapy is typically not used. This is because radiation to the entire lining of the lung has many side effects that are often severe including damage to the lung (pneumonitis). There is a new radiation technique using Intensity Modulated Radiation Therapy (IMRT) that has been shown to reduce many of the side effects of standard radiation therapy. This type of radiation therapy specifically targets the lining of the lung, where you have your cancer, and reduces the risk of damaging the lung itself. The purpose of this study is to test the safety and implementation of standard pleurectomy/decortication (removal of the surface lining of the lung) and standard chemotherapy followed by IMRT performed at other centers. Patients will undergo pleurectomy/decortication chemotherapy and hemithoracic pleural IMRT to the pleura in patients with malignant pleural mesothelioma.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent to participate on the study
* Patients must have a pathologically confirmed diagnosis either at MSKCC or at the participating site of stage I-III malignant pleural mesothelioma
* Epithelioid or biphasic histology subtype (Note: patients with biphasic histology can have < 10% sarcomatoid)
* No evidence of metastatic disease.
* Patient age ≥ 18 years but ≤ 80 years at the time of consent.
* Karnofsky performance status ≥ 80%
* Pulmonary Function Tests:

  1. For all patients: DLCO > 40% predicted (corrected for Hgb)
  2. For patients enrolled post-P/D, only: FEV1 >/= 35% (corrected for Hgb) (Note: patients enrolled prior to P/D will have PFTs repeated pre-IMRT. If this criteria is not met, they will be removed from study)
* In cases of concern about decreased renal function and potential high radiation dose to the kidneys, an optional nuclear medicine kidney function scan may be performed prior to radiation therapy to determine the functional contribution of each kidney.
* Patient enrolled prior to chemotherapy must have adequate organ function as indicated by the following laboratory values:

  1. Absolute neutrophil count ≥1.5 K/mcL
  2. Platelets ≥100 K/mcL
  3. Serum total bilirubin ≤ 1.5 X ULN
  4. AST (SGOT) or ALT (SGPT) ≤ 3.0 X ULN Note: patients enrolled after chemotherapy do not have to meet the above criteria

Exclusion Criteria:

* > 10% Sarcomatoid or desmoplastic histology
* Continuous oxygen use
* Prior nephrectomy on the contralateral side of MPM
* Prior intrapleural therapy (except pleurodesis) or intrapleural therapy at the time of P/D (i.e.: intrapleural chemotherapy, photodynamic therapy, intrapleural betadine)
* Prior thoracic radiation therapy preventing hemithoracic pleural IMRT
* Bulky disease in the fissure preventing lung-sparing pleural IMRT
* Patients undergoing extrapleural pneumonectomy
* Patients with an active infection that require systemic antibiotics, antiviral, or antifungal treatments
* Patients with a concurrent active malignancy (except squamous or basal cell carcinoma of the skin)
* Patients with serious unstable medical illness
* Presence of third space fluid that cannot be controlled by drainage
* For patients who develop or have baseline clinically significant pleural effusions before or during initiation of pemetrexed therapy; consideration should be given to drain the effusion prior to chemotherapy administration
* No acute congestive heart failure
* Pregnant or lactating women
* Men or women not using effective contraception

Reproductive risks Patients should not become pregnant or father a baby while on this study because the drugs in this study can affect an unborn baby. Women should not breast-feed a baby while on this study. Women of childbearing age will be counseled to use birth control while on this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-10-11; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
number of patients ≥ grade 3 pneumonitis | 2 years
  Grade 3 pneumonitis is defined as symptomatic, interfering with ADL's and requiring oxygen support as defined by the NCI Common Terminology Criteria (CTC) version 4.0 for toxicity and Adverse Event reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Simone, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (12):
- United States (12):
  - Moffitt Cancer Center, Tampa, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack, Commack, New York
  - Memoral Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Rockville Center, NY, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Md Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Rimner A, Zauderer MG, Gomez DR, Adusumilli PS, Parhar PK, Wu AJ, Woo KM, Shen R, Ginsberg MS, Yorke ED, Rice DC, Tsao AS, Rosenzweig KE, Rusch VW, Krug LM. Phase II Study of Hemithoracic Intensity-Modulated Pleural Radiation Therapy (IMPRINT) As Part of Lung-Sparing Multimodality Therapy in Patients With Malignant Pleural Mesothelioma. J Clin Oncol. 2016 Aug 10;34(23):2761-8. doi: 10.1200/JCO.2016.67.2675. Epub 2016 Jun 20. PMID 27325859
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org